CLINICAL TRIAL: NCT05136027
Title: Exercise Program in Patients With Treatment-resistant Depressive Disorder Compared to Usual Practice
Brief Title: TReAtment With CombinedExercise in Patients With Resistant Major Depression
Acronym: TRACE-RMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Collaborators: Red Salud Mental Araba (Other Government)
Responsible Party: Principal Investigator, SARA MALDONADO-MARTIN, Head of laboratory, Principal Investigator, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRACE-RMD study
Record Dates: First submitted 2021-11-01; First posted 2021-11-26 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Resistant Depression, Treatment
Keywords: Depression; Exercise; Low-intensity Interval Training; Resistance Training
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression; Motor Activity

STUDY DESIGN:
Intervention Model Description: Exercise group Atenttion Control
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group: In the exercise session will carry out a combined training in four parts, low- intensity interval training in a bicycle, resistance circuit training, low- intensity interval training in a bicycle, and CORE exercises.
  Interventions: Other: Combined training
- Attention Control (No Intervention): Regular in-hospital treatment with occupational activity sessions with the same frequency and duration as the intervention group.

INTERVENTIONS:
Other: Combined training — Low-intensity interval training and resistance exercise
  Arms: Intervention group

SUMMARY:
Major depressive disorder is one of the most prevalent and disabling mental disorders worldwide. Forty percent of people with major depressive disorder are in moderate remission, with the remainder meeting the criteria for treatment-resistant depressive disorder (TRD), with an inadequate response to at least two different antidepressants of adequate dose and duration. Dysfunctionality in these individuals is frequent and severe and its importance contrasts with the absence of drugs to alleviate these deficits. Exercise programs, which were initially developed as interventions aimed at improving physical health in early stages or in mild symptomatology, have shown that they can also improve the symptoms of this disease in more advanced stages There is evidence of new therapeutic interventions for TRD. New pharmacological targets that aim to improve the evolution of depression and its functional repercussions augur that, in the future, new drugs will have to be combined with other therapeutic strategies, including exercise. Therefore, the objectives of this clinical trial with a control group are: 1) to analyze the changes in depressive symptoms in people diagnosed with TRD included in the exercise program compared to a control group; 2) to evaluate the improvement in physical health through cardiovascular risk factors and life expectancy suffered by this sector of the population, and 3) to analyze changes in functional status and quality of life. This is a prospective longitudinal intervention design (three months) in which people with TRD are included in two groups: 1) intervention with exercise (two days/week) and 2) control care with usual treatment. The aim is to find an improvement in mood and functionality with the implementation of exercise, as well as changes in physical areas such as blood pressure or body mass index, which are considered predictive factors of cardiovascular disease.

DETAILED DESCRIPTION:
The presence of major depressive disorder (MDD) in today's society is worryingly high. Specifically, the prevalence-year prevalence of MDD in Spain is 3.9% and lifetime prevalence is 10.5%. The lifetime prevalence for men is 6.29% and 14.47% for women in Spain according to the ESEMED-Spain study. Although there is no explicit international consensus, the medical literature and research define treatment-resistant depression (TRD) as any MDD that does not respond to two trials of treatment antidepressant treatment at adequate doses and for an adequate duration of time.

MDD is the leading cause of years lived with disability worldwide, accounting for 11.9%. It has been estimated that during the year 2020 it could be second only to ischemic heart disease in disability-adjusted life years lost. Given this bleak scenario, different non-pharmacological strategies have been considered as possible complementary treatments to pharmacological treatment to help improve the prognosis of MDD and remission rates, such as exercise and electroconvulsive therapy.

Sedentary lifestyles are a very common feature in the severely mentally disordered population. One of the causes for this to occur is that people with MDD have very little confidence in their ability to exercise and lack the necessary social support. This inactivity together with other modifiable risk factors such as tobacco use, high blood pressure, and overweight/obesity, in addition to the side effects of pharmacological treatments contributes to the appearance of different diseases, as well as decreased life expectancy and quality of life. TRD can act as a cause or as a repercussion of physical inactivity.

It has been recognized for several years that the performance of regular exercise is cardioprotective, decreasing the incidence of cardiovascular diseases such as arterial hypertension, coronary artery disease, type 2 diabetes, and atherosclerosis. In addition to being cardioprotective, exercise has shown a positive association with psychological well-being and therapeutic benefits in older people with depressive disorder, depressive symptoms in patients with Alzheimer's disease and MDD.

Although there is still some controversy about the intensity and frequency of exercise, and the duration of the exercise program, the recommendations were the adoption of a moderate-intensity exercise program of at least 30 minutes on most days of the week, for 10-12 weeks. In the latest World Health Organization guidelines on physical activity (PA) and sedentary habits, for the improvement of quality of life in adults with TMD the general recommendations do not differ from the general population, i.e., people should accumulate throughout the week a minimum of 150-300 minutes of moderate aerobic PA or a minimum of 75-150 minutes of vigorous PA, or an equivalent combination of both in order to obtain notable health benefits. Also, in order to achieve additional health benefits, the participants should perform two days a week of moderate or higher intensity muscle-strengthening activities.

ELIGIBILITY:
Inclusion Criteria:

* Depression major disorder.
* 2 or more antdepressives resistant a treatment.
* Consent informed signed

Exclusion Criteria:

* Schizophrenia or other disorders.
* Suicide risk.
* Unstable medic illness or unsuitable controlled.
* Disorder for use of active substances.
* Comorbidity with other psychiatric pathologies.
* Montreal Cognitive Assessment <26/30, cognitive deterioration.
* Incapacity for realizing physical exercise because of osteoarticular, cardiovascular, or metabolic difficulty.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depressión Rating Scale (MADRS) | 12 weeks
  Ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders.
  Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
  Usual cutoff points are:
  0 to 6 - normal /symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression
Cardiorespiratory fitness | 12 weeks
  Cardiorespiratory fitness evaluation measured by cardiopulmonary exercise test. Maximu oxygen uptake measured in mL/kg/min or L/min is the gold standard variable.

SECONDARY OUTCOMES:
Clinical Global Impression Scale (CGI) | 12 weeks
  The Clinical Global Impression (CGI) rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders. Its 3 items assess, 1) Severity of Illness (CGI-S), 2) Global Improvement (CGI-I), and 3) Efficacy Index (CGI-E, which is a measure of treatment effect and side effects specific to drugs that were administered).
Sheehan Disability Scale (SDS) | 12 weeks
  five-item, self-rated questionnaire designed to measure the extent to which a patient's disability due to an illness or health problem interferes with work/school, social life/leisure activities, and family life/home responsibilities.
  Total score 0-30 (0 unimpaired, 30 highly impaired) Work/school (0-10) Social life (0-10) Family life/home responsibilities (0-10 Scores of ≥5 on any of the 3 scales; high scores are associated with significant functional impairment.
Treatment Satisfaction Questionnaire for Medication - 9 items (TSQM-9) | 12 weeks
  To measure patients' satisfaction with medication

CONTACTS AND LOCATIONS:
Overall Officials: NAGORE IRIARTE-YOLLER, MD, Principal Investigator — PSYCHIATRIC HOSPITAL OF ÁLAVA
Locations (1):
- Basque Country University, Vitoria-Gasteiz, Spain

IPD SHARING:
Plan to Share IPD: Yes
A protocol paper will be written once the clinical trials identification number will be defined
Supporting Information: Study Protocol
Time Frame: indefinite period
Access Criteria: no criteria

REFERENCES:
- [Derived] Tous-Espelosin M, Pavon-Navajas C, Etxaniz-Oses J, Canas-Garcia MT, Maldonado-Martin S, Orruno-Vivar J, Corres P, Iriarte-Yoller N. Effects of combined exercise training for adults with resistant major depression: a pilot study from the TRACE-RMD project. PeerJ. 2025 Nov 17;13:e20356. doi: 10.7717/peerj.20356. eCollection 2025. PMID 41282982
- [Derived] Iriarte-Yoller N, Etxaniz-Oses J, Pavon-Navajas C, Tous-Espelosin M, Sanchez-Gomez PM, Maldonado-Martin S, Yoller-Elburgo AB, Elizagarate-Zabala E. Treatment with combined exercise in patients with resistant major depression (TRACE-RMD): study protocol for a randomised controlled trial. Trials. 2024 Dec 18;25(1):827. doi: 10.1186/s13063-024-08685-7. PMID 39696604